CLINICAL TRIAL: NCT01881165
Title: A Randomized, Double-blind, Placebo Controlled Trial Evaluating the Effectiveness of a Cranberry Concentrate in Preventing Recurrent Urinary Tract Infections in Adult Women
Brief Title: Cranberry on Urinary Tract Infections
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor declined funding
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H13-01491
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cranberry (Experimental): Each capsule contains 500 mg of cranberry powder at a concentration ratio of 36:1 (36 grams of cranberries equals 1 gram of concentrate).
  Interventions: Drug: Cranberry
- Placebo (Placebo Comparator): A capsule containing control formulation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cranberry
  Arms: Cranberry
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study aims to determine whether a cranberry concentrate reduces recurrent urinary tract infections (UTIs) in women who consume it. About 150 adult women will participate in this study. Subjects will be randomized (like flipping a coin) to take either cranberry capsule or a placebo for 12 months. We expect cranberry supplement to have better results than the placebo. Subjects will not know which supplement they are taking. The primary outcome is the number of UTIs over 12 months.

DETAILED DESCRIPTION:
Participants will attend their first study visit at a clinic at UBC. They will be randomized to the cranberry capsule or placebo. Participants will be instructed to consume the assigned supplement for the next 12 months. A calendar will be provided to record compliance and recurrent UTI. Participants will also record any side effects. They will be phoned each month to encourage participation and adherence. At 8 weeks and 6 months, they will be asked to return to the clinic to complete a midline questionnaire which will ask about any recurrent UTIs experienced. More supplements will be provided at their 6-month visit. At 12 months, participants will return to the clinic to complete an endline questionnaire. They will return any leftover supplements, calendar and side effect diary. If participants withdraw from the study, they will still be encouraged to return at 12 months to complete the survey to allow for intent-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Females who have had at least 2 clinical-diagnosed symptomatic UTIs in the year preceding
* Are sexually active

Exclusion Criteria:

* Current UTI
* Pregnant or breastfeeding or planning a pregnancy in the next 12 months
* A known allergy or intolerance to cranberry-containing products
* A history of renal stones and/or renal transplantation
* Any immunosuppressive disease or other medical conditions that could potentially interfere with outcomes
* Current use of corticosteroid, anticoagulant, antidepressants or mood stabilizing medications or other medications that may interact with the supplement
* Intermittent or indwelling catheterization
* Any anatomic abnormalities of the urinary tract
* The use of any antibiotics within 2 weeks before study entry
* The use of any natural health products, including herbs, homeopathic products, or other forms of cranberry supplements within 2 weeks before study entry

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Number of urinary tract infections | 12 months
  The number of symptomatic UTIs over 12 months (defined by self-report as having one or more of the following symptoms: dysuria, frequency, urgency, hematuria, supra-pubic pressure or fever), the proportion of participants with at least 1 symptomatic UTI, the median time to the first UTI

SECONDARY OUTCOMES:
Side effects | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tim Green, PhD, Principal Investigator — University of British Columbia
Locations (1):
- The University of British Columbia, Vancouver, British Columbia, Canada